CLINICAL TRIAL: NCT06358898
Title: Effect of a Smartphone-based, Mood-enhanced Cognitive Behavioral Therapy for Insomnia in Adolescents At Risk of Depression: A Cluster Randomized Trial
Brief Title: Digital Mood-enhanced CBT-I to Improve Depressive Symptoms in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN NGAN YIN, Assistant Professor, Department of Psychiatry, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20221207
Record Dates: First submitted 2024-04-02; First posted 2024-04-11 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Depression; Adolescent
Keywords: Insomnia; Depression; Adolescent
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard dCBT-I (Active Comparator): Treatment content for insomnia was structured and based on the well-established CBT elements for treating insomnia, with developmental adaptation and age-appropriate modification specific for adolescent population. For example, regularity of sleep wake pattern and circadian component will be further emphasized in this age group given the high prevalence of social jetlag resulting from the early school schedule and their natural development delay in circadian rhythm.
  Interventions: Behavioral: Standard dCBT-I
- Modified Mood enhanced CBT-I (M-dCBT-I) (Experimental): For mood-enhanced dCBT-I (M-dCBT-I), apart from including core CBT-I component, additional depression specific component including behavioral activation and problem solving. More specifically, cognitive restructuring techniques will cover both unhelpful belief relevant to both insomnia and depression. Psychoeducation will also cover both condition and vignette example will be included in the treatment.
  Interventions: Behavioral: Modified Mood enhanced CBT-I (M-dCBT-I)

INTERVENTIONS:
Behavioral: Standard dCBT-I — This standard digital CBT-I intervention will cover (1) psycho-education about sleep, circadian and sleep hygiene education, (2) stimulus control, (3) sleep restriction, (4) relaxation techniques, (5) structured worry time, (6) cognitive restructuring (targeting sleep-related dysfunctional cognitions), and (7) relapse prevention. In order to have comparable dosage as modified CBT-I, the treatment will be dispersed to 8 modules (8-week) which is still in the range of standard CBT-I duration (usually last for 6-8weeks).
  Arms: Standard dCBT-I
Behavioral: Modified Mood enhanced CBT-I (M-dCBT-I) — Additional depression specific components will be added to the standard CBT-I, including behavioral activation and problem solving.
  Arms: Modified Mood enhanced CBT-I (M-dCBT-I)

SUMMARY:
Emerging encouraging evidence showed that sleep focused treatment can simultaneously improve sleep and depression in adult with comorbid conditions. Although these favorable changes in depressed adults is encouraging, little is known in the potential efficacy of CBT-I in altering depression trajectory in adolescent population. This current study aims to compare the effect of digitally delivered, mood enhanced cognitive behavioral therapy for insomnia (M-dCBT-I) and standard digital cognitive behavioral therapy for insomnia (dCBT-I) in improving depressive symptoms in adolescents, and to examine the potential sustained treatment effect in mood outcomes following M-dCBT-I or dCBT-I treatment.

DETAILED DESCRIPTION:
Adolescence is a critical transitional stage accompanied by the emergence of mental disorders, with major depressive disorder (MDD) being the most common mental disorder. The point prevalence of depression ranges from 3% to 18% across different studies. In addition, according to our previous studies, approximately 10% of adolescents experience insomnia disorders, and 36% have insomnia symptoms. Adolescent concurrently experiencing sleep and mood problems are typically at a higher risk of adverse health outcomes. This particular group is usually much more difficult to treat, with a poorer prognosis, suggesting that this group maybe in particular need for effective treatment.

There is accumulating evidence that adolescent sleep and mood problems can be treated successfully using cognitive behavioral therapy (CBT), which is one of the most extensively evaluated non-pharmacological approach for managing either depression or insomnia symptoms in adolescents. Cognitive behavioral therapy for depression (CBT-D) involves psychoeducation and addresses cognitive restructuring for unrealistic thinking contribute to depressed mood and behavioral strategies to increase pleasant activities. While cognitive behavioral therapy for insomnia (CBT-I) is the first-line treatment in managing adult insomnia, it has gained increasing empirical evidence in managing adolescent insomnia. The high comorbidity of insomnia and depression calls for the need for addressing both problems due to the fact that residual insomnia or residual depressive symptoms could further hasten a relapse to the other comorbid disorder. In addition, depression becomes more difficult to treat in the presence of insomnia. In fact, there has, however, been emerging encouraging evidence showing that sleep focused treatment can simultaneously improve sleep and depression in adult with comorbid conditions. Although these favorable changes in depressed adults is encouraging, little is known in the potential efficacy of CBT-I in altering depression trajectory in adolescent population.

This current study aims to compare the effect of digitally delivered, mood enhanced cognitive behavioral therapy for insomnia (M-dCBT-I) and standard digital cognitive behavioral therapy for insomnia (dCBT-I) in improving depressive symptoms in adolescents, and to examine the potential sustained treatment effect in mood outcomes following M-dCBT-I or dCBT-I treatment. Primary outcomes include the depressive symptoms as measured by PHQ-9, while secondary outcomes include clinician rated depression scale (HRSD), insomnia (ISI), sleep-related measures (Sleep diary variables, dysfunctional sleep belief), daytime sleepiness, anxiety (HADS), quality of life (Kidscreen-27). Outcome measurement will be conducted at baseline, postintervention, 6-month and 12-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adolescent aged 12-18 years old
2. presence of insomnia problems as defined by insomnia severity index ≥ 9 (locally validated cut off for detecting clinical insomnia in adolescents)
3. presence of depressive problems as defined by Patient Health Questionnaire-9 (PHQ-9) using cut off of 10 for detecting clinical depression
4. ability to read and understand Chinese
5. possession of smartphone

Exclusion Criteria:

1. presence of prominent suicidality (suicide plans and suicide attempts) as determined by the Mini-International Neuropsychiatric Interview (MINI)
2. a clinical diagnosis of psychosis, schizophrenia, bipolar disorders, or intellectual disability
3. presence of other sleep disorders that significantly affect sleep continuity or sleep quality (e.g. restless leg symptoms or obstructive sleep apnea syndrome) as determined by validated Diagnostic Interview for Sleep Patterns and Disorders
4. currently receiving psychological treatment for insomnia and/or pharmacological treatment for depression

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 343 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  The severity of depressive symptoms as measured by Patient Health Questionnaire 9-item (PHQ-9): locally validated in adolescents and commonly used self-administered questionnaire to assess depressive symptoms and severity. Scores range from 0 to 27, with higher score indicate higher level of depression.

SECONDARY OUTCOMES:
Assessor-rated depressive symptomatology | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Hamilton Rating Scale for Depression (HRSD), a 17-item clinician-administered instrument, will be used to assess depressive symptomatology. Scores range from 0 to 52, with higher score indicate higher level of depression.
Overall severity of depression symptoms | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Improvement of depression, in reference to the severity prior to the start of the treatment, will be rated using the Clinical Global Improvement Scale (CGI-I), on a scale of 1 (very much improved) to 7 (very much worse).
Severity of insomnia symptoms | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Severity of insomnia symptoms will be measured by Insomnia Severity Index (ISI). ISI is a self-report measure designed to assess the nature, severity and impact of insomnia, with a higher total score suggesting more severe insomnia symptoms. Scores range from 0 to 28.
Sleep-wake pattern | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Prospective 7-day Sleep diary will be used to record sleep-wake pattern including sleep duration, wakeup time, bedtime and sleep latency.
Sleep-related beliefs and cognitions | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) will be used to measure faulty sleep-related beliefs and cognitions, which are cognitive aspects typically involved in the maintenance of insomnia. The total score is calculated from the average score of all the items on the scale and could range from 0 to 10.
Daytime sleepiness | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  8-item Pediatric Daytime Sleepiness Scale (PDSS) will be used to assess adolescents' daytime sleepiness in school children and adolescents. It is an 8-item inventory designed for use with school children and youths, with a higher score indicating greater sleepiness. Scores ranged from 0 to 32.
Anxiety and depression symptoms | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Cantonese-Chinese version Hospital Anxiety and Depression Scale (HADS) will be used to assess anxiety and depression. It has been validated in the community-based sample of adolescents in Hong Kong.
  A higher total score of each subscale represents a greater severity of depression/anxiety. The total score for each subscale ranges from 0 to 21.
Quality of life by KIDSCREEN-27 | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  KIDSCREEN-27 health questionnaire for children and young people will be used to measure quality of life.
  A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.

OTHER OUTCOMES:
Major life events and self-perceived stress | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Life Experience Survey (LES) will be used to measure major life events and self-perceived stress associated with these events that an individual experienced over the year.
Chronotype | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Morningness-Eveningness Questionnaire (MEQ) will be used to measure the chronotype of the study participants.
  Individuals scored higher than 17 and lower than 12 were classified as morning-type and evening-type, respectively. Individuals scored between 12 and 17 were classified as intermediate-type. Scores range from 4 to 25.
Pubertal status | Baseline, Postintervention (8 weeks), 6-month follow up and 12-month follow up
  Self-rated tanner stage will be used to measure pubertal status of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Ngan Yin Chan, PhD, Principal Investigator — Department of Psychiatry, the Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, the Chinese University of Hong Kong, Shatin, New Territories, Hong Kong